CLINICAL TRIAL: NCT04686760
Title: Efficacy of Inhaled Nitroglycerin in Moderate to Severe Cases of COVID-19 Patients
Brief Title: Efficacy of Inhaled Nitroglycerin in Moderate to Critically Ill COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Mansoor Hafeez, Doctor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBEC/BIH/08-2020
Record Dates: First submitted 2020-12-24; First posted 2020-12-29 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitroglycerin solution (Experimental)
  Interventions: Drug: Nitroglycerin
- standard solution (No Intervention)

INTERVENTIONS:
Drug: Nitroglycerin — 2 mg/ml solution of nitroglycerin used for nebulization four hourly
  Arms: Nitroglycerin solution

SUMMARY:
In current analysis moderate to severely ill Covid-19 infected patients will be nebulized with nitroglycerin, and they will be compared with the standard nebulization

ELIGIBILITY:
Inclusion Criteria:

Diagnosed admitted cases of Covid-19 degree of illness should be moderate to severe both male and female every age group

Exclusion Criteria:

allergic to nitroglycerin sudden drop in blood pressure not given consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
ratio of partial pressure of oxygen in arterial blood to fraction of inhaled oxygen | 5-7 days
Oxygen demand | 5-7 days

SECONDARY OUTCOMES:
Duration of hospital stay | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria Town International Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided